CLINICAL TRIAL: NCT00304629
Title: Long Term Safety and Efficacy of Galantamine in Alzheimer's Disease (Extension INT-8)
Brief Title: Long-term Safety and Efficacy of Galantamine in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012070
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; cholinesterase inhibitors; galantamine
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine

SUMMARY:
The long-term safety and efficacy of galantamine (12 mg bid) will be documented during a one year open-label treatment in subjects with Alzheimer's Disease who completed the GAL-INT-8 trial (up to 400 eligible patients). Safety will be tracked by means of adverse event reports, laboratory parameters and physical exam. Long-term efficacy will be evaluated by means of a Alzheimer's Disease Assessment Scale(ADAS) and activities of daily living scale Disability Assessment for Dementia Scale(DAD)

DETAILED DESCRIPTION:
This is a twelve-month, open-label trial in which treatment with 12 mg bid galantamine will be evaluated. Only subjects who took trial medication during the 24-month trial period of GAL-INT-8 will be eligible. Safety will be assessed by periodic physical examination, vital signs, ECG and laboratory tests and reports of adverse events. The ADAS-cognitive scale and DAD scale will be used to document long-term efficacy.

Patients will be seen at 6 monthly intervals but the ADAS-cognitive scale and DAD scale will only be performed at end of trial. The treatment will consist of tablets which will contain 12 mg of galantamine. Duration of treatment equals 12 months. Patients will receive 1 tablet twice daily preferably to be taken with food (breakfast in the morning at approximately 8 AM and a snack or meal in the evening at approximately 6PM).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have taken trial medication during the 24-month trial period of GAL-INT-8 and should be enrolled within 1 month after completion
* Patients and their primary caregiver give informed consent for the participation in the trial
* Patients must have remained in good health, as determined by medical history, complete physical examination and laboratory tests

Exclusion Criteria:

* If a patient developed, during the trial GAL-INT-8, symptoms of other neurological or psychiatric diseases that might contribute to dementia, the subject cannot be enrolled. This includes subjects developing neurodegenerative disorders such as Parkinson's disease, Pick's disease or Huntington's chorea, or Creutzfeldt-Jacob disease, and subjects with cognitive impairment resulting from stroke, acute cerebral trauma, hypoxic cerebral damage, infection or primary or metastatic cerebral neoplasia
* Subjects with the following co-existing medical conditions: a) Any history of epilepsy or convulsions except for febrile convulsions during childhood b) Peptic ulcer: if the ulcer is considered to be still "active", i.e., if treatment for this condition started <3 months ago or if treatment is not successful (symptoms still present), the subject is not eligible. c) Clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances
* Patients with current, clinically significant cardiovascular disease that would be expected to limit the subject's ability to complete a 12-month trial. The following would usually be considered clinically significant cardiovascular disease: a) Unstable angina
* angina or coronary artery disease that required a change in medication (anti-angina or digitalis) within the last 3 months b) Decompensated congestive heart failure i.e. when symptoms occur in a subject on stable medication during rest or light exercise (NYHA III and IV). Note: if the only signs of decompensation are pretibial or malleolar oedema and the exercise tolerance is still reasonable (absence of dyspnoea) the subject should not be excluded c) Cardiac disease potentially resulting in syncope, near syncope or other alterations of mental status
* In addition, the following conditions should lead to exclusion: atrial fibrillation without prophylactic treatment to prevent thromboembolic stroke, bradycardia <50 beats/min., atrioventricular block > first degree. d) Severe mitral or aortic valvular disease e) Hypotension or treatment for hypotension f) Systolic blood pressure greater than 170 mmHg or diastolic blood pressure greater than 110 mmHg
* Patients using any agent for the treatment of dementia (approved, experimental, including over the counter agents), including, but not limited to nootropic agents, cholinomimetic agents, choline, oestrogens taken without medical need, chronic NSAIDs (30 consecutive days), vitamin E more than 30 IU daily, and deprenyl
* Conditions that could interfere with the absorption of the compound or with the evaluation of the disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2000-03; Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is safety as measured by adverse events, laboratory tests, vital signs, weight, physical exam and electrocardiogram

SECONDARY OUTCOMES:
The secondary outcome is effectiveness as measured by a cognitive scale (ADAS) and by activities of daily living (DAD).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] Rockwood K, Dai D, Mitnitski A. Patterns of decline and evidence of subgroups in patients with Alzheimer's disease taking galantamine for up to 48 months. Int J Geriatr Psychiatry. 2008 Feb;23(2):207-14. doi: 10.1002/gps.1864. PMID 17621382